CLINICAL TRIAL: NCT00436748
Title: A Multi-Center, Double-Blind, Randomized Study Evaluating De Novo Weekly and Once Every Two Week Darbepoetin Alfa Dosing for the Correction of Anemia in Pediatric Subjects With Chronic Kidney Disease Receiving and Not Receiving Dialysis
Brief Title: Study to Assess Darbepoetin Alfa Dosing for the Correction of Anemia in Pediatric Patients With Chronic Kidney Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA and EMA agreed that the information that had been submitted to date was acceptable to meet the requirements of the post-marketing commitment.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20050256
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Anemia; Chronic Kidney Disease; Kidney Disease
Keywords: Chronic Kidney Disease; Dialysis; Anemia; Nephrology; Pediatric; Hemodialysis; Peritoneal Dialysis; Chronic Renal Insufficiency
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Diseases | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darbepoetin Alfa QW (Experimental): Participants received darbepoetin alfa once a week (QW) for 24 weeks. The initial dose was 0.45 μg/kg; thereafter, active doses were administered to achieve and then maintain hemoglobin levels within a target range of 10.0 to 12.0 g/dL. Participants not on dialysis or who were receiving peritoneal dialysis were administered darbepoetin alfa subcutaneously; participants receiving hemodialysis were administered darbepoetin alfa intravenously.
  Interventions: Drug: Darbepoetin Alfa
- Darbepoetin Alfa Q2W (Experimental): Participants received darbepoetin alfa every 2 weeks (Q2W) and a placebo every other 2 weeks to maintain the blind for 24 weeks. The initial dose was 0.75 μg/kg; thereafter, active doses were administered to achieve and then maintain hemoglobin levels within a target range of 10.0 to 12.0 g/dL. Participants not on dialysis or who were receiving peritoneal dialysis were administered darbepoetin alfa subcutaneously; participants receiving hemodialysis were administered darbepoetin alfa intravenously.
  Interventions: Drug: Darbepoetin Alfa; Drug: Placebo

INTERVENTIONS:
Drug: Darbepoetin Alfa — Administered by subcutaneous or intravenous injection
  Other Names: Aranesp®
Drug: Placebo — Matching placebo solution for subcutaneous or intravenous injection to maintain the blind in the Q2W arm.
  Arms: Darbepoetin Alfa Q2W

SUMMARY:
The primary objectives of this study are the following:

1. To test if the proportion of participants achieving a hemoglobin value greater than or equal to 10.0 g/dL at any time point after the first dose during the study is greater than 0.8 when administered de novo darbepoetin alfa once a week (QW) for treatment of anemia in pediatric patients with chronic kidney disease receiving and not receiving dialysis, and
2. To test if the proportion of participants achieving a hemoglobin value greater than or equal to 10.0 g/dL at any time point after the first dose during the study is greater than 0.8 when administered de novo darbepoetin alfa every 2 weeks (Q2W) for treatment of anemia in pediatric patients with chronic kidney disease receiving and not receiving dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Chronic Kidney Disease, either receiving or not receiving dialysis
* Anemic, with two consecutive screening hemoglobin values drawn at least 7 days apart < 11.0 g/dL
* Transferrin saturation (Tsat) greater than or equal to 20%

Exclusion Criteria:

* Any erythropoiesis stimulating agent (ESA) use within 12 weeks prior to randomization
* other hematologic disorders
* upper or lower gastrointenstinal bleeding within 6 months prior to randomization
* uncontrolled hypertension
* prior history (within 12 weeks prior to randomization) of acute myocardial ischemia, hospitalization for congestive heart failure, myocardial infarction, stroke or transient ischemic attack
* prior history (within 6 months prior to randomization) of thromboembolism

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2008-09-16 (Actual); Primary Completion 2014-03-03 (Actual); Study Completion 2014-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (63):
- United States (39):
  - Research Site, Birmingham, Alabama
  - Research Site, Los Angeles, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Kansas City, Missouri
  - Research Site, Livingston, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Valhalla, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Ghent
  - Research Site, Leuven
- Research Site, Jūrmala, Latvia
- Research Site, Vilnius, Lithuania
- Mexico (4):
  - Research Site, Mexico City, Mexico City
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Puebla City
- Poland (3):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Szczecin
- Research Site, San Juan, Puerto Rico
- Russia (5):
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Orenburg
  - Research Site, Saint Petersburg
  - Research Site, Samara
- Slovakia (3):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
- United Kingdom (3):
  - Research Site, Birmingham
  - Research Site, Leeds
  - Research Site, London

REFERENCES:
- [Background] Warady BA, Barcia J, Benador N, Jankauskiene A, Olson K, Podracka L, Shavkin A, Srivaths P, Wong CJ, Petersen J. De novo weekly and biweekly darbepoetin alfa dosing in pediatric patients with chronic kidney disease. Pediatr Nephrol. 2018 Jan;33(1):125-137. doi: 10.1007/s00467-017-3758-5. Epub 2017 Aug 17. PMID 28815341
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial enrolled pediatric patients with chronic kidney disease (CKD) who were anemic and not treated with an erythropoiesis-stimulating agent (ESA). The study was conducted at 43 centers in the US, Europe and Mexico. The first participant was enrolled on 16 September 2008 and the last participant was enrolled on 02 December 2013.
Pre-assignment Details: A total of 189 participants were screened, 116 participants were enrolled, and 73 screen failed. The primary reasons for screen failure were hemoglobin concentration > 10 g/dL or transferrin saturation < 20%. Randomization was stratified by age and dialysis status.
Period: Overall Study
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Started | 59 | 57
Received Treatment | 58 | 56
Completed | 48 | 45
Not Completed | 11 | 12
Not completed — Ineligibility Determined | 1 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Consent Withdrawn | 1 | 4
Not completed — Administrative Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol-specified Criteria | 5 | 4
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Population: Efficacy analysis set, including all participants who received ≥ 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W | Total
Number analyzed (Participants) | 58 | 56 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (3.6) | 12.8 (3.7) | 12.7 (3.6)
Age, Customized [Number; unit: participants]
  1 - < 6 years | 2 | 1 | 3
  6 - < 12 years | 19 | 18 | 37
  12 - 18 years | 37 | 37 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 35 | 33 | 68
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 30 | 30 | 60
  Black or African American | 4 | 5 | 9
  Hispanic or Latino | 23 | 20 | 43
  Other | 1 | 1 | 2
Dialysis Status [Number; unit: participants]
  Not receiving dialysis | 33 | 33 | 66
  Receiving hemodialysis | 15 | 14 | 29
  Receiving peritoneal dialysis | 10 | 9 | 19
Hemoglobin Concentration [Mean (Standard Deviation); unit: g/dL] | 8.59 (0.84) | 8.73 (0.84) | 8.66 (0.84)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving Hemoglobin ≥ 10.0 g/dL
Description: The proportion of participants achieving hemoglobin ≥ 10.0 g/dL (the correction proportion) was calculated as the number of participants achieving a hemoglobin ≥ 10.0 g/dL at any time point during the study when administered de novo darbepoetin alfa without receiving any red blood cell transfusion after randomization and within 90 days before the achievement, divided by the number of participants in the efficacy analysis set.
Time Frame: 24 weeks
Population: Efficacy analysis set
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 58 | 56
proportion of participants | 0.983 [0.908 to 1.000] | 0.839 [0.717 to 0.924]
Statistical Analysis 1: Comparison: Darbepoetin Alfa QW; The null hypothesis for the Darbepoetin Alfa QW group was that the correction proportion (p) ≤ 0.8 ; Th alternative hypothesis was that p > 0.8. The correction proportion was compared with 0.8 using the exact method to test the null hypothesis at a 1-sided overall significance level of 0.025; Test type: Superiority or Other; p < 0.001, Exact
Statistical Analysis 2: Comparison: Darbepoetin Alfa Q2W; The null hypothesis for the Darbepoetin Alfa Q2W group was that the correction proportion (p) ≤ 0.8 ; Th alternative hypothesis was that p > 0.8. The correction proportion was compared with 0.8 using the exact method to test the null hypothesis at a 1-sided overall significance level of 0.025; Test type: Superiority or Other; p = 0.293, Exact

2. Secondary Outcome: Time to First Hemoglobin Value ≥ 10.0 g/dL
Description: The time from study Day 1 to the day a participant first achieved hemoglobin ≥ 10.0 g/dL for participants who achieved hemoglobin ≥ 10.0 g/dL.
Time Frame: 24 weeks
Population: Efficacy analysis set responders (participants with at least 1 postbaseline hemoglobin ≥ 10.0 g/dL)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 57 | 47
days | 24.0 [15.0 to 50.0] | 22.0 [14.0 to 41.0]

3. Secondary Outcome: Hemoglobin Concentration Over Time
Time Frame: Baseline and Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24 and 25.
Population: Efficacy analyis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 58 | 56
g/dL
  Baseline (n=58, 56) | 8.59 (0.84) | 8.73 (0.84)
  Week 1 (n=53, 50) | 8.64 (0.90) | 8.65 (0.95)
  Week 2 (n=52, 52) | 8.74 (1.09) | 8.96 (1.20)
  Week 3 (n=51, 55) | 9.28 (1.27) | 9.09 (1.27)
  Week 4 (n=53, 53) | 9.79 (1.30) | 9.55 (1.23)
  Week 5 (n=53, 52) | 10.18 (1.29) | 9.87 (1.32)
  Week 6 (n=54, 50) | 10.54 (1.43) | 10.19 (1.33)
  Week 7 (n=52, 48) | 10.96 (1.53) | 10.17 (1.25)
  Week 8 (n=53, 51) | 11.05 (1.37) | 10.47 (1.21)
  Week 9 (n=50, 51) | 11.03 (1.48) | 10.60 (1.34)
  Week 10 (n=54, 51) | 11.32 (1.33) | 10.60 (1.29)
  Week 11 (n=51, 48) | 11.34 (1.33) | 10.73 (1.22)
  Week 12 (n=51, 48) | 11.45 (1.25) | 10.87 (1.38)
  Week 13 (n=50, 47) | 11.68 (1.19) | 10.82 (1.33)
  Week 14 (n=52, 50) | 11.27 (1.28) | 10.92 (1.31)
  Week 15 (n=49, 50) | 11.25 (1.13) | 11.00 (1.23)
  Week 16 (n=48, 47) | 11.36 (1.19) | 10.86 (1.21)
  Week 17 (n=48, 48) | 11.21 (1.23) | 11.05 (1.00)
  Week 18 (n=49, 46) | 11.14 (1.20) | 10.91 (1.09)
  Week 19 (n=48, 46) | 11.06 (0.91) | 10.91 (1.09)
  Week 20 (n=48, 45) | 11.09 (1.03) | 10.76 (1.00)
  Week 21 (n=48, 46) | 11.20 (1.04) | 10.64 (0.99)
  Week 22 (n=48, 45) | 11.00 (1.19) | 10.58 (1.04)
  Week 23 (n=48, 44) | 10.93 (1.10) | 10.50 (1.05)
  Week 24 (n=45, 46) | 10.93 (1.16) | 10.43 (0.97)
  Week 25 (n= 32, 31) | 11.13 (1.10) | 10.65 (0.75)

4. Secondary Outcome: Weight-adjusted Darbepoetin Alfa Dose at Time of Achieving First Hemoglobin ≥ 10.0 g/dL
Description: The darbepoetin alfa dose at the time a participant achieved a first hemoglobin level ≥ 10.0 g/dL, divided by the participant's weight measured at the closest study week prior to the dosing, post dialysis.
Time Frame: 24 weeks
Population: Efficacy analysis set responders (participants with at least 1 postbaseline hemoglobin ≥ 10.0 g/dL) for whom dosing data were available.
Measure: Mean (Standard Deviation); unit: μg/kg
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 54 | 44
μg/kg | 0.48 (0.24) | 0.76 (0.21)

5. Secondary Outcome: Darbepoetin Alfa Weight-Adjusted Dose Over Time
Description: Arithmetic means are provided; Withheld doses are counted as 0 μg.
Time Frame: Day 1 (initial dose) and Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24 and 25.
Population: Efficacy analyis set with available data at each time point (indicated by "n"). Numbers > 0 on non-darbepoetin alfa dosing weeks for the Q2W group reflect participants who did not receive the assigned placebo dose (eg, dose withheld per investigator decision based on hemoglobin value or missed visit).
Measure: Mean (Standard Deviation); unit: μg/kg
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 58 | 56
μg/kg
  Initial Dose (n=58, 56) | 0.45 (0.07) | 0.73 (0.13)
  Week 2 (n=55, 0) | 0.45 (0.07) | NA (NA) — Participants received dosing every 2 weeks
  Week 3 (n=55, 52) | 0.44 (0.07) | 0.72 (0.11)
  Week 4 (n=54, 0) | 0.40 (0.11) | NA (NA) — Participants received dosing every 2 weeks
  Week 5 (n=54, 51) | 0.43 (0.26) | 0.72 (0.25)
  Week 6 (n=54, 0) | 0.42 (0.29) | NA (NA) — Participants received dosing every 2 weeks
  Week 7 (n=54, 51) | 0.38 (0.25) | 0.70 (0.28)
  Week 8 (n=53, 1) | 0.34 (0.24) | 0.00 (NA) — Could not be calculated since sample size = 1
  Week 9 (n=52, 52) | 0.32 (0.23) | 0.64 (0.26)
  Week 10 (n=55, 3) | 0.33 (0.26) | 0.00 (0.00)
  Week 11 (n=54, 50) | 0.32 (0.28) | 0.61 (0.35)
  Week 12 (n=54, 2) | 0.26 (0.28) | 0.00 (0.00)
  Week 13 (n=54, 50) | 0.24 (0.28) | 0.56 (0.35)
  Week 14 (n=53, 4) | 0.21 (0.27) | 0.00 (0.00)
  Week 15 (n=52, 48) | 0.31 (0.33) | 0.53 (0.36)
  Week 16 (n=50, 5) | 0.35 (0.44) | 0.00 (0.00)
  Week 17 (n=51, 47) | 0.29 (0.34) | 0.61 (0.97)
  Week 18 (n=50, 3) | 0.32 (0.40) | 0.00 (0.00)
  Week 19 (n=50, 46) | 0.31 (0.33) | 0.45 (0.30)
  Week 20 (n=48, 4) | 0.35 (0.34) | 0.00 (0.00)
  Week 21 (n=48, 46) | 0.38 (0.63) | 0.47 (0.36)
  Week 22 (n=48, 3) | 0.38 (0.64) | 0.00 (0.00)
  Week 23 (n=47, 44) | 0.39 (0.63) | 0.49 (0.40)
  Week 24 (n=46, 1) | 0.41 (0.63) | 0.00 (NA) — Could not be calculated since sample size = 1

6. Secondary Outcome: Change From Baseline at Week 13 and Week 25 in Parent-reported Pediatric Quality of Life Inventory (PedsQL) Scores
Description: The PedsQL is a health-related quality of life (HRQOL) questionnaire that can be used to measure quality of life in children ≥ 2 years old. The 23-item PedsQL 4.0 includes physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), and school functioning (5 items). Separate questionnaires for ages 2 to 4 (toddler), 5-7, 8-12, and 13-18 years are used for parent proxy-reporting, which assesses parents' perceptions of their child's HRQOL. The instructions ask how much of a problem each item has been during the past 1 month; each item is answered on a 5-point scale: 0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem. Scores from the 4 subscales, the total score, and the psychosocial composite score were generated using standard algorithms. Each item's score in the questionnaire was converted to a 0 to 100 scale (with higher scores indicating better HRQOL).
Time Frame: Baseline, Week 13 and Week 25 (or end of study visit if earlier than Week 25)
Population: Efficacy analysis set with available data for each score at each time point (indicated by "n").
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 45 | 46
units on a scale
  Week 13 Total Score (n=45, 46) | 4.50 (2.19) | 0.58 (2.43)
  Week 13 Psychosocial composite score (n=45, 46) | 5.12 (2.16) | -0.41 (2.57)
  Week 13 Physical function score (n=45, 46) | 3.61 (3.20) | 2.31 (3.35)
  Week 13 Emotional function score (n=45, 46) | 1.00 (3.00) | -3.89 (2.74)
  Week 13 Social function score (n=45, 46) | 6.89 (3.54) | 0.76 (3.56)
  Week 13 School function score (n=42, 42) | 7.30 (2.47) | 4.17 (3.63)
  Week 25 Total Score (n=38, 41) | 1.90 (2.06) | 0.65 (2.66)
  Week 25 Psychosocial composite score (n=38, 41) | 2.52 (1.83) | -1.84 (3.13)
  Week 25 Physical function score (n=38, 41) | 0.66 (3.89) | 5.18 (3.59)
  Week 25 Emotional function score (n=38, 41) | -0.66 (2.61) | -3.51 (3.16)
  Week 25 Social function score (n=38, 41) | 5.13 (2.64) | -2.20 (4.10)
  Week 25 School function score (n=36, 37) | 3.90 (2.51) | 2.03 (3.94)

7. Secondary Outcome: Change From Baseline at Week 13 and Week 25 in Child Self-reported Pediatric Quality of Life Inventory (PedsQL) Scores
Description: The PedsQL child self-reported questionnaire was used in children > 5 years old. The 23-item PedsQL 4.0 includes physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), and school functioning (5 items). Separate questionnaires for ages 5-7, 8-12, and 13-18 years was used for child self-reporting. The instructions asked how much of a problem each item has been during the past 1 month; each item is answered on a 5-point scale for ages 8 to 18 (0 = never a problem; 1 = almost never a problem; 2 = sometimes a problem; 3 = often a problem; 4 = almost always a problem), or simplified to a 3-point scale for ages 5 to 7 (0 = not at all a problem; 2 = sometimes a problem; 4 = a lot of a problem). Scores from the 4 subscales, the total score, and the psychosocial composite score were generated using standard algorithms. Each item's score in the questionnaire was converted to a 0 to 100 scale (with higher scores indicating better HRQOL).
Time Frame: Baseline, Week 13 and Week 25 (or end of study visit if earlier than Week 25)
Population: Efficacy analysis set aged > 5 years and with available data for each score at each time point (indicated by "n").
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 46 | 46
units on a scale
  Week 13 Total Score (n=46, 46) | 2.94 (1.70) | -1.23 (2.04)
  Week 13 Psychosocial composite score (n=46, 46) | 2.59 (1.92) | -0.45 (2.23)
  Week 13 Physical function score (n=46, 46) | 3.78 (2.43) | -2.79 (2.59)
  Week 13 Emotional function score (n=46, 46) | 0.43 (2.52) | -0.76 (2.79)
  Week 13 Social function score (n=46, 46) | 3.26 (2.93) | -2.28 (3.02)
  Week 13 School function score (n=45, 43) | 2.89 (2.98) | 2.44 (3.83)
  Week 25 Total Score (n=40, 42) | 5.00 (1.75) | 2.58 (1.78)
  Week 25 Psychosocial composite score (n=40, 42) | 3.81 (1.97) | 3.53 (2.01)
  Week 25 Physical function score (n=40, 42) | 7.42 (2.48) | 0.74 (2.80)
  Week 25 Emotional function score (n=40, 42) | -0.25 (2.51) | 3.93 (3.10)
  Week 25 Social function score (n=40, 42) | 7.00 (3.10) | 2.50 (2.67)
  Week 25 School function score (n=40, 39) | 4.25 (3.14) | 3.85 (3.09)

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: A serious adverse event (SAE) is defined as an adverse event that meets at least one of the following serious criteria: • is fatal, • is life threatening, • requires in-patient hospitalization or prolongation of existing hospitalization, • results in persistent or significant disability/incapacity, • is a congenital anomaly/birth defect, and/or • other significant medical hazard. The investigator assessed whether the adverse event was related to the investigational product (IP). Events of interest included hypertension, ischemic heart disease, cardiac failure, cerebrovascular disorders, convulsions, embolic and thrombotic events, embolic and thrombotic events: venous, embolic and thrombotic events: arterial, embolic and thrombotic events: vessel type unspecified and mixed arterial and venous, dialysis vascular access thrombosis, antibody-mediated pure red cell aplasia, hypersensitivity, lack of efficacy-effect, and malignancies.
Time Frame: 25 weeks
Population: Safety analysis set including all participants who received ≥ 1 dose of investigational product.
Measure: Number; unit: participants
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 58 | 56
participants
  All adverse events | 48 | 50
  Serious adverse events | 16 | 14
  Leading to discontinuation of IP | 0 | 2
  Leading to discontinuation from study | 0 | 2
  Fatal adverse events | 0 | 0
  Events of interest | 18 | 20
  Treatment-related adverse events (TRAE) | 14 | 16
  Treatment-related serious adverse events | 1 | 2
  TRAE leading to discontinuation of IP | 0 | 2
  TRAE leading to discontinuation from study | 0 | 2
  Treatment-related fatal adverse events | 0 | 0
  Treatment-related events of interest | 6 | 9

9. Secondary Outcome: Hemoglobin Serial Rate of Change (ROC) Over Time
Description: Calculated using the serial method as the change in hemoglobin from the previous non-missing hemoglobin level divided by number of days in between, and then multiplied by 7.
Time Frame: Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24 and 25.
Population: Safety analyis set with available data at each time point (indicated by "n").
Measure: Median (Full Range); unit: g/dL/week
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 58 | 56
g/dL/week
  Week 2 (n=49, 47) | 0.263 (1.09) [-0.90 to 1.17] | 0.350 (1.20) [-1.82 to 2.10]
  Week 3 (n=50, 53) | 0.530 (1.27) [-1.00 to 1.70] | 0.200 (1.27) [-1.23 to 1.40]
  Week 4 (n=53, 52) | 0.560 (1.30) [-0.40 to 2.20] | 0.513 (1.23) [-1.60 to 3.33]
  Week 5 (n=53, 49) | 0.438 (1.29) [-2.00 to 2.00] | 0.117 (1.32) [-3.92 to 1.52]
  Week 6 (n=54, 48) | 0.400 (1.43) [-2.50 to 2.40] | 0.231 (1.33) [-1.05 to 2.40]
  Week 7 (n=51, 45) | 0.200 (1.53) [-1.20 to 2.90] | 0.100 (1.25) [-1.75 to 2.57]
  Week 8 (n=52, 49) | 0.163 (1.37) [-1.98 to 1.63] | 0.300 (1.21) [-2.71 to 1.17]
  Week 9 (n=49, 50) | 0.100 (1.48) [-2.80 to 1.40] | 0.089 (1.34) [-1.30 to 2.20]
  Week 10 (n=53, 50) | 0.117 (1.33) [-1.40 to 3.90] | 0.000 (1.29) [-2.10 to 1.52]
  Week 11 (n=51, 48) | 0.100 (1.33) [-2.10 to 1.87] | 0.138 (1.22) [-1.49 to 1.49]
  Week 12 (n=51, 48) | 0.000 (1.25) [-1.40 to 4.40] | 0.200 (1.38) [-2.20 to 1.10]
  Week 13 (n=50, 47) | 0.128 (1.19) [-2.80 to 2.70] | -0.064 (1.33) [-2.57 to 2.19]
  Week 14 (n=52, 50) | -0.419 (1.28) [-1.87 to 2.40] | 0.023 (1.31) [-1.40 to 1.40]
  Week 15 (n=49, 50) | 0.200 (1.13) [-1.60 to 2.33] | 0.128 (1.23) [-2.38 to 1.63]
  Week 16 (n=48, 47) | 0.000 (1.19) [-2.10 to 3.27] | -0.100 (1.21) [-3.20 to 1.10]
  Week 17 (n=47, 48) | -0.100 (1.23) [-2.80 to 2.40] | 0.139 (1.00) [-1.00 to 2.00]
  Week 18 (n=48, 46) | -0.188 (1.20) [-2.30 to 1.40] | 0.094 (1.09) [-2.33 to 1.40]
  Week 19 (n=47, 46) | 0.100 (0.91) [-1.52 to 1.20] | -0.100 (1.09) [-2.22 to 3.90]
  Week 20 (n=47, 44) | 0.000 (1.03) [-1.90 to 2.60] | -0.050 (1.00) [-3.20 to 1.10]
  Week 21 (n=47, 45) | 0.100 (1.04) [-1.48 to 2.45] | -0.140 (0.99) [-1.20 to 1.40]
  Week 22 (n=48, 44) | -0.200 (1.19) [-2.60 to 1.10] | 0.000 (1.04) [-1.70 to 1.60]
  Week 23 (n=47, 43) | -0.100 (1.10) [-2.80 to 1.75] | 0.000 (1.05) [-1.54 to 1.82]
  Week 24 (n=44, 46) | 0.100 (1.16) [-3.03 to 4.34] | 0.050 (0.97) [-1.60 to 6.44]
  Week 25 (n=32, 31) | 0.188 (1.10) [-1.20 to 2.10] | 0.000 (0.75) [-1.05 to 1.68]

10. Secondary Outcome: Number of Participants With Hemoglobin > 12.0, > 13.0, and > 14.0 g/dL During the Study
Time Frame: 25 weeks
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 58 | 56
participants
  Number of participants with hemoglobin > 12.0 g/dL | 44 | 33
  Number of participants with hemoglobin > 13.0 g/dL | 24 | 6
  Number of participants with hemoglobin > 14.0 g/dL | 6 | 2

11. Secondary Outcome: Maximum Increase in Hemoglobin Over Any 2 Week Period
Description: The maximum increase between any 2 non-missing hemoglobin measurements over any 2-week period from Day 1.
Time Frame: 25 weeks
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: g/dL/2 weeks
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 58 | 56
g/dL/2 weeks | 2.06 (0.88) | 1.61 (0.76)

12. Secondary Outcome: Change From Baseline in Systolic Blood Pressure Over Time
Time Frame: Baseline and Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24 and 25.
Population: Safety analyis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 58 | 56
mmHg
  Week 2 (n=55, 54) | 1.7 (11.6) [-0.90 to 1.17] | -3.9 (11.1) [-1.82 to 2.10]
  Week 3 (n=55, 56) | 1.1 (14.1) [-1.00 to 1.70] | 0.0 (12.7) [-1.23 to 1.40]
  Week 4 (n=55, 54) | 1.3 (13.0) [-0.40 to 2.20] | 1.2 (11.5) [-1.60 to 3.33]
  Week 5 (n=55, 52) | 1.1 (13.7) [-2.00 to 2.00] | -3.0 (13.7) [-3.92 to 1.52]
  Week 6 (n=54, 51) | 0.2 (14.2) [-2.50 to 2.40] | -2.9 (12.5) [-1.05 to 2.40]
  Week 7 (n=54, 52) | -1.0 (14.2) [-1.20 to 2.90] | -3.7 (13.4) [-1.75 to 2.57]
  Week 8 (n=55, 52) | 0.5 (16.0) [-1.98 to 1.63] | -2.7 (13.8) [-2.71 to 1.17]
  Week 9 (n=54, 52) | 1.0 (18.3) [-2.80 to 1.40] | -3.1 (14.5) [-1.30 to 2.20]
  Week 10 (n=55, 52) | -0.2 (16.6) [-1.40 to 3.90] | -3.7 (14.6) [-2.10 to 1.52]
  Week 11 (n=54, 51) | -2.0 (15.6) [-2.10 to 1.87] | -1.8 (15.9) [-1.49 to 1.49]
  Week 12 (n=55, 49) | -2.4 (17.2) [-1.40 to 4.40] | -2.8 (15.4) [-2.20 to 1.10]
  Week 13 (n=53, 50) | 0.5 (14.8) [-2.80 to 2.70] | -2.1 (14.2) [-2.57 to 2.19]
  Week 14 (n=54, 50) | -2.3 (19.5) [-1.87 to 2.40] | -1.8 (15.8) [-1.40 to 1.40]
  Week 15 (n=53, 50) | 0.1 (17.4) [-1.60 to 2.33] | -2.4 (13.0) [-2.38 to 1.63]
  Week 16 (n=50, 48) | 1.9 (16.4) [-2.10 to 3.27] | -3.8 (16.3) [-3.20 to 1.10]
  Week 17 (n=51, 47) | 1.0 (17.7) [-2.80 to 2.40] | 0.1 (10.6) [-1.00 to 2.00]
  Week 18 (n=50, 46) | 0.5 (18.5) [-2.30 to 1.40] | 0.0 (15.5) [-2.33 to 1.40]
  Week 19 (n=50, 47) | 3.4 (16.0) [-1.52 to 1.20] | -2.5 (14.2) [-2.22 to 3.90]
  Week 20 (n=48, 46) | -0.9 (18.3) [-1.90 to 2.60] | -4.0 (13.0) [-3.20 to 1.10]
  Week 21 (n=49, 46) | 1.9 (15.7) [-1.48 to 2.45] | -2.2 (15.0) [-1.20 to 1.40]
  Week 22 (n=48, 46) | -0.6 (18.2) [-2.60 to 1.10] | -0.9 (15.0) [-1.70 to 1.60]
  Week 23 (n=47, 45) | -0.6 (16.5) [-2.80 to 1.75] | -1.2 (15.7) [-1.54 to 1.82]
  Week 24 (n=46, 46) | 0.0 (17.8) [-3.03 to 4.34] | -2.0 (11.8) [-1.60 to 6.44]
  Week 25 (n=34, 32) | -0.5 (14.3) [-1.20 to 2.10] | -2.3 (12.4) [-1.05 to 1.68]

13. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure Over Time
Time Frame: Baseline and Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24 and 25.
Population: Safety analyis set with available data at each time point (indicated by "n").
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 58 | 56
mmHg
  Week 2 (n=55, 54) | 1.4 (9.4) [-0.90 to 1.17] | 0.8 (11.1) [-1.82 to 2.10]
  Week 3 (n=55, 56) | 2.2 (11.0) [-1.00 to 1.70] | 3.1 (10.8) [-1.23 to 1.40]
  Week 4 (n=55, 54) | 2.8 (11.0) [-0.40 to 2.20] | 1.8 (12.6) [-1.60 to 3.33]
  Week 5 (n=55, 52) | 3.0 (12.4) [-2.00 to 2.00] | -0.2 (11.2) [-3.92 to 1.52]
  Week 6 (n=54, 51) | 2.6 (10.1) [-2.50 to 2.40] | -0.1 (11.4) [-1.05 to 2.40]
  Week 7 (n=54, 52) | 1.2 (10.4) [-1.20 to 2.90] | -1.0 (12.3) [-1.75 to 2.57]
  Week 8 (n=55, 52) | 3.9 (11.9) [-1.98 to 1.63] | 1.1 (15.0) [-2.71 to 1.17]
  Week 9 (n=54, 52) | 4.8 (14.7) [-2.80 to 1.40] | -0.3 (12.9) [-1.30 to 2.20]
  Week 10 (n=55, 52) | 1.5 (13.7) [-1.40 to 3.90] | 0.9 (15.9) [-2.10 to 1.52]
  Week 11 (n=54, 51) | 3.9 (11.8) [-2.10 to 1.87] | 0.9 (14.4) [-1.49 to 1.49]
  Week 12 (n=55, 49) | 1.6 (10.4) [-1.40 to 4.40] | 2.8 (13.7) [-2.20 to 1.10]
  Week 13 (n=54, 50) | 2.7 (13.8) [-2.80 to 2.70] | 2.2 (10.6) [-2.57 to 2.19]
  Week 14 (n=54, 50) | 3.4 (14.4) [-1.87 to 2.40] | 1.7 (12.0) [-1.40 to 1.40]
  Week 15 (n=53, 50) | 3.7 (12.9) [-1.60 to 2.33] | 1.4 (11.7) [-2.38 to 1.63]
  Week 16 (n=50, 48) | 4.6 (13.7) [-2.10 to 3.27] | 0.7 (11.9) [-3.20 to 1.10]
  Week 17 (n=51, 47) | 4.1 (15.6) [-2.80 to 2.40] | 2.6 (10.6) [-1.00 to 2.00]
  Week 18 (n=50, 46) | 3.0 (16.4) [-2.30 to 1.40] | 0.4 (11.7) [-2.33 to 1.40]
  Week 19 (n=50, 47) | 3.7 (12.9) [-1.52 to 1.20] | 0.6 (12.2) [-2.22 to 3.90]
  Week 20 (n=48, 46) | 1.7 (13.8) [-1.90 to 2.60] | 2.0 (13.2) [-3.20 to 1.10]
  Week 21 (n=49, 46) | 2.9 (15.1) [-1.48 to 2.45] | 0.6 (12.9) [-1.20 to 1.40]
  Week 22 (n=48, 46) | 3.2 (14.7) [-2.60 to 1.10] | 0.3 (13.9) [-1.70 to 1.60]
  Week 23 (n=47, 45) | 5.0 (13.8) [-2.80 to 1.75] | -2.0 (14.0) [-1.54 to 1.82]
  Week 24 (n=46, 46) | 4.0 (13.8) [-3.03 to 4.34] | -0.3 (12.8) [-1.60 to 6.44]
  Week 25 (n=34, 32) | 3.0 (13.0) [-1.20 to 2.10] | -1.5 (10.7) [-1.05 to 1.68]

14. Secondary Outcome: Number of Participants Who Developed Anti-erythropoiesis Antibodies
Description: Participants who were negative for anti-erythropoiesis antibodies at Baseline (pre-dose) and who developed anti-erythropoiesis antibodies during the study. Serum samples were tested using Amgen's Surface Plasmon Resonance Immunoassay (SPRIA) method.
Time Frame: 25 weeks
Population: Safety analysis set with both pre and postdose immunoassay antibody results
Measure: Number; unit: participants
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 49 | 49
participants | 2 | 4

15. Secondary Outcome: Darbepoetin Alfa Serum Concentrations for Participants Less Than 6 Years of Age
Description: Serum concentrations of darbepoetin alfa were measured by an enzyme-linked immunosorbent assay (ELISA).
Time Frame: Weeks 1, 2, and 3 before the investigational product dose and 2 days after the first investigational product dose
Population: Due to the low number of participants <6 years of age summary concentration analyses were not performed.
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 25 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Darbepoetin Alfa QW | Darbepoetin Alfa Q2W
Serious Adverse Events (participants affected / at risk) | 16/58 | 14/56
Other Adverse Events (participants affected / at risk) | 42/58 | 43/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa QW (N=58) | Darbepoetin Alfa Q2W (N=56)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Device failure (General disorders) | 1 | 0
Device malfunction (General disorders) | 1 | 1
Local swelling (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 1
Oedema (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 2
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Shunt infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Gastrostomy failure (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 2 | 0
Vesical fistula (Renal and urinary disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 3
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Darbepoetin Alfa QW (N=58) | Darbepoetin Alfa Q2W (N=56)
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 4 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 10 | 9
Catheter site pain (General disorders) | 3 | 1
Fatigue (General disorders) | 5 | 2
Injection site pain (General disorders) | 3 | 2
Medical device complication (General disorders) | 2 | 3
Pyrexia (General disorders) | 5 | 10
Catheter site infection (Infections and infestations) | 4 | 3
Ear infection (Infections and infestations) | 4 | 0
Nasopharyngitis (Infections and infestations) | 4 | 6
Pharyngitis (Infections and infestations) | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 7
Urinary tract infection (Infections and infestations) | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3
Procedural hypotension (Injury, poisoning and procedural complications) | 3 | 3
Blood pressure increased (Investigations) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Dizziness (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 4 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Hypertension (Vascular disorders) | 9 | 8
Hypotension (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.